CLINICAL TRIAL: NCT00204282
Title: The Effectiveness of Nurse Practitioner Led Group Visits in Improving Compliance With Diabetic Preventative Services and Modifying Vascular Risk
Brief Title: The Effectiveness of Improving Compliance With Diabetic Preventative Services and Modifying Vascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 12567A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes
Keywords: Diabetes prevention
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surveys and Questionnaires

INTERVENTIONS:
Behavioral: Educational presentation, group discussion, questionnaires

SUMMARY:
The purpose of the study is to evaluate the feasibility and efficacy of group visits led by nurse practitioners in improving diabetic preventive services and vascular risk. Diabetes is notable for its high burden on the health of urban populations, a rich literature supporting evidenced based care, and great opportunities to apply systemic primary care interventions to reduce its toll. Extensive literature demonstrates sub-optimal care in the community as well as in academic centers. Addressing the needs of patients with diabetes is challenging in the primary-care environment and nurse case management and disease-specific group visits which focus on education and self-management skills have been shown to be useful adjuncts to traditional outpatient care.

The study will attempt to demonstrate that nurse practitioner run group visits, during which the NP will provide didactic education, facilitate group interaction, and arrange referrals and laboratory testing as appropriate, will improve compliance with established American Diabetes Association guidelines for screening and preventive care and in doing so lower cardiovascular risk. Satisfaction with care, quality of life, and diabetic knowledge will be assessed before and after the patients complete the program. In addition, we will attempt to characterize barriers to care for patients who were formerly established with a primary care physician in the Primary Care Group, but who have not received diabetic care there for at least one year.

DETAILED DESCRIPTION:
Patients who are 40 to 79 years old, and who have had at least three visits with a primary care physician will be the focus of the study. Patients will be recruited by letter, co-signed by the PCP and the study P1 A second letter will be sent 2 weeks after the first. After an intake visit, random allocation will divide 150 patients into 2 arms, one a series of 3 NP-led group classes and the other, usual care. Baseline data, including blood pressure control, foot and retinal examination rates, serum lipids, Alc, microalbumin, pneumococcal vaccination, smoking status and counseling, and ASA and lipid medication use will be assessed at enrollment and again at completion of the study. In addition patients will complete a diabetic knowledge scale, quality of life assessment (SF- 12) and ADA patient satisfaction survey. Several measures will be gathered both by chart review and oral administration of the CDC's BRFSS 2002 diabetes module survey, permitting cross validation. Statistical analysis of the differences between proportions (2x2 for independent samples) will be performed using chi-square. Preliminary power analysis (Power Precision; Biostat, Englewood, NJ) suggests adequate power (using Fisher's exact test, alpha beta 0.1, assuming reasonably achievable effect sizes) for at least several intermediate outcomes.

Patients in the 'group visit' arm are expected to attend three 90-minute educational group visits over six months, with group visits directed by a nurse practitioner. Patients will be asked to attend three sessions (8-10 patients in each) within six months. All patients will continue to see their primary care physicians as scheduled. The focus of the visits will be on diabetic and vascular risk goals, dietary education, and self-management skills. A graphical 'Diabetic Health Tracker' modified from Chapin et al will be provided to group class attendees; such an intervention may improve vascular risk endpoints. The group visit provider team will have the ability to make referrals, administer recommended vaccines, and adjust medications in consultation with the primary care physician; NPs will also make phone contact with the class group members between visits to report results and help assure follow-up; such case management functions may also improve outcomes. Additional telephone outreach will be made to patients who both: 1) do respond to the 2 recruiting letters, and 2) who have not been seen in the past 12 months in order review barriers to care. A brief phone screen for depression will be considered given data linking depression to non-adherence.

As the burden of chronic illness rises along with healthcare costs, innovative approaches are required. Diabetes care has been repeatedly identified by government and private payers as area of focus and perhaps even a future subject for "pay for performance". We hope our study can contribute to better diabetic care and, in the longer term, to improved patient health.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients age 40-79 who are followed in the Primary Care Group for Type 2 diabetes and who have seen their PCP at least 3 times in order to establish regular care

Exclusion Criteria:

* Patients younger than 40 years of age

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-08; Study Completion 2005-12

PRIMARY OUTCOMES:
Nurse practitioner run group visits will improve compliance with established American Diabetes Association guidelines for screening and preventive care

SECONDARY OUTCOMES:
Compliance with established American Diabetes Association guidelines for screening and preventive care will lower cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davis, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Saydah SH, Eberhardt MS, Loria CM, Brancati FL. Age and the burden of death attributable to diabetes in the United States. Am J Epidemiol. 2002 Oct 15;156(8):714-9. doi: 10.1093/aje/kwf111. PMID 12370159
- [Background] Institute of Medicine (US) Committee on Identifying Priority Areas for Quality Improvement; Adams K, Corrigan JM, editors. Priority Areas for National Action: Transforming Health Care Quality. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK221294/ PMID 25057643
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Adler AI, Stratton IM, Neil HA, Yudkin JS, Matthews DR, Cull CA, Wright AD, Turner RC, Holman RR. Association of systolic blood pressure with macrovascular and microvascular complications of type 2 diabetes (UKPDS 36): prospective observational study. BMJ. 2000 Aug 12;321(7258):412-9. doi: 10.1136/bmj.321.7258.412. PMID 10938049
- [Background] American Diabetes Association: clinical practice recommendations. Standards of medical for patients with diabetes mellitus. Diabetes Care 2003; 26:(suppl 1):533-50
- [Background] Fleming BB, Greenfield S, Engelgau MM, Pogach LM, Clauser SB, Parrott MA. The Diabetes Quality Improvement Project: moving science into health policy to gain an edge on the diabetes epidemic. Diabetes Care. 2001 Oct;24(10):1815-20. doi: 10.2337/diacare.24.10.1815. No abstract available. PMID 11574448
- [Background] Centers for Disease Control and Prevention (CDC). Preventive-care practices among persons with diabetes--United States, 1995 and 2001. MMWR Morb Mortal Wkly Rep. 2002 Nov 1;51(43):965-9. PMID 12433019
- [Background] Saaddine JB, Engelgau MM, Beckles GL, Gregg EW, Thompson TJ, Narayan KM. A diabetes report card for the United States: quality of care in the 1990s. Ann Intern Med. 2002 Apr 16;136(8):565-74. doi: 10.7326/0003-4819-136-8-200204160-00005. PMID 11955024
- [Background] Grant RW, Cagliero E, Murphy-Sheehy P, Singer DE, Nathan DM, Meigs JB. Comparison of hyperglycemia, hypertension, and hypercholesterolemia management in patients with type 2 diabetes. Am J Med. 2002 Jun 1;112(8):603-9. doi: 10.1016/s0002-9343(02)01103-8. PMID 12034408
- [Background] Sobel BE, Frye R, Detre KM; Bypass Angioplasty Revascularization Investigation 2 Diabetes Trial. Burgeoning dilemmas in the management of diabetes and cardiovascular disease: rationale for the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Trial. Circulation. 2003 Feb 4;107(4):636-42. doi: 10.1161/01.cir.0000048897.03553.e4. PMID 12566379
- [Background] Chin MH, Zhang JX, Merrell K. Diabetes in the African-American Medicare population. Morbidity, quality of care, and resource utilization. Diabetes Care. 1998 Jul;21(7):1090-5. doi: 10.2337/diacare.21.7.1090. PMID 9653601
- [Background] Renders CM, Valk GD, Griffin SJ, Wagner EH, Eijk Van JT, Assendelft WJ. Interventions to improve the management of diabetes in primary care, outpatient, and community settings: a systematic review. Diabetes Care. 2001 Oct;24(10):1821-33. doi: 10.2337/diacare.24.10.1821. PMID 11574449
- [Background] Sadur CN, Moline N, Costa M, Michalik D, Mendlowitz D, Roller S, Watson R, Swain BE, Selby JV, Javorski WC. Diabetes management in a health maintenance organization. Efficacy of care management using cluster visits. Diabetes Care. 1999 Dec;22(12):2011-7. doi: 10.2337/diacare.22.12.2011. PMID 10587835
- [Background] Norris SL, Nichols PJ, Caspersen CJ, Glasgow RE, Engelgau MM, Jack L, Isham G, Snyder SR, Carande-Kulis VG, Garfield S, Briss P, McCulloch D. The effectiveness of disease and case management for people with diabetes. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):15-38. doi: 10.1016/s0749-3797(02)00423-3. PMID 11985933
- [Background] Montori VM, Dinneen SF, Gorman CA, Zimmerman BR, Rizza RA, Bjornsen SS, Green EM, Bryant SC, Smith SA; Translation Project Investigator Group. The impact of planned care and a diabetes electronic management system on community-based diabetes care: the Mayo Health System Diabetes Translation Project. Diabetes Care. 2002 Nov;25(11):1952-7. doi: 10.2337/diacare.25.11.1952. PMID 12401738
- [Background] Olivarius NF, Beck-Nielsen H, Andreasen AH, Horder M, Pedersen PA. Randomised controlled trial of structured personal care of type 2 diabetes mellitus. BMJ. 2001 Oct 27;323(7319):970-5. doi: 10.1136/bmj.323.7319.970. PMID 11679387
- [Background] Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med. 2003 Jan 30;348(5):383-93. doi: 10.1056/NEJMoa021778. PMID 12556541
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Vrijhoef HJ, Diederiks JP, Spreeuwenberg C, Wolffenbuttel BH, van Wilderen LJ. The nurse specialist as main care-provider for patients with type 2 diabetes in a primary care setting: effects on patient outcomes. Int J Nurs Stud. 2002 May;39(4):441-51. doi: 10.1016/s0020-7489(01)00046-3. PMID 11909620
- [Background] Lenz ER, Mundinger MO, Hopkins SC, Lin SX, Smolowitz JL. Diabetes care processes and outcomes in patients treated by nurse practitioners or physicians. Diabetes Educ. 2002 Jul-Aug;28(4):590-8. doi: 10.1177/014572170202800413. PMID 12224199
- [Background] Rickheim PL, Weaver TW, Flader JL, Kendall DM. Assessment of group versus individual diabetes education: a randomized study. Diabetes Care. 2002 Feb;25(2):269-74. doi: 10.2337/diacare.25.2.269. PMID 11815494
- [Background] Chapin RB, Williams DC, Adair RF. Diabetes control improved when inner-city patients received graphic feedback about glycosylated hemoglobin levels. J Gen Intern Med. 2003 Feb;18(2):120-4. doi: 10.1046/j.1525-1497.2003.20367.x. PMID 12542586
- [Background] Rachmani R, Levi Z, Slavachevski I, Avin M, Ravid M. Teaching patients to monitor their risk factors retards the progression of vascular complications in high-risk patients with Type 2 diabetes mellitus--a randomized prospective study. Diabet Med. 2002 May;19(5):385-92. doi: 10.1046/j.1464-5491.2002.00701.x. PMID 12027926
- [Background] Ciechanowski PS, Katon WJ, Russo JE. Depression and diabetes: impact of depressive symptoms on adherence, function, and costs. Arch Intern Med. 2000 Nov 27;160(21):3278-85. doi: 10.1001/archinte.160.21.3278. PMID 11088090
- [Background] Terry K. Better quality care, bigger paycheck. Med Econ. 2002 Sep 9;79(17):99-100, 103-6, 109-10. No abstract available. PMID 12298136
- [Background] Hawryluk M: CMS project to measure physician quality of care. Am Med News. American Medical Association. February 2003